CLINICAL TRIAL: NCT07049328
Title: A Phase 1 Study of HCW9302, an IL-2 Fusion Protein, for Alopecia Areata
Brief Title: HCW9302 (Interleukin-2 Fusion Protein) for Alopecia Areata
Acronym: IL-2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HCW Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCWALO101
Record Dates: First submitted 2025-06-04; First posted 2025-07-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-08

CONDITIONS: Alopecia Areata(AA)
Keywords: Alopecia; Interleukin-2 (IL-2); T-Reg
MeSH Terms: conditions — Alopecia Areata; Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study of HCW9302, an IL-2 fusion protein, for alopecia areata (Experimental): Single dose subcutaneous injection of HCW9302.
  Interventions: Drug: HCW9302, an IL-2 fusion protein

INTERVENTIONS:
Drug: HCW9302, an IL-2 fusion protein — Injection

SUMMARY:
This is a Phase 1, open-label, multi-center, competitive enrollment, and dose-escalation study of HCW9302 in subjects with Alopecia Areata (AA)

DETAILED DESCRIPTION:
The study involves dose escalation to determine the toxicity profile of HCW9302 and to designate a dose level for the Phase 2 expansion phase (RP2D).

Up to five HCW9302 dose levels will be evaluated. A step-down dose level (level -1) will be provided in the event that unacceptable toxicity is encountered at the planned initial dose level. In the first stage of the study, HCW9302 will be administered subcutaneously as a single dose. Depending on the results of the single ascending dose stage, a multidose study of HCW9302 administered subcutaneously every 28 days for 4 consecutive treatments will be considered.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women who are 18 to 70 years of age, or adult males who are 18 to 60 years of age at the time of informed consent.
2. Clinical diagnosis of Alopecia Areata (AA) (including ophiasis, totalis or universalis forms) at Screening.
3. Negative serum pregnancy test within 14 days of treatment start if female and of childbearing potential (non-childbearing is defined as greater than one year postmenopausal or surgically sterilized).
4. Female subjects of childbearing potential must adhere to using a highly effective medically accepted method of birth control (defined as those with failure less than 1%; see Appendix 2) prior to screening and agree to continue its use for at least 28 days after the last dose of HCW9302 or be surgically sterilized (e.g., hysterectomy or tubal ligation) and males must agree to use a barrier method of birth control and agree to continue its use for at least 28 days after the last dose of HCW9302.
5. Laboratory tests performed within 28 days of treatment start:

   1. Absolute neutrophil count (AGC/ANC) ≥ 1,500/μL (≥1.5 × 109/L)
   2. Platelets ≥ 100,000/μL (≥ 100 × 109/L)
   3. Hemoglobin ≥ 10 g/dL (>100g/L)
   4. Calculated glomerular filtration rate (GFR)* >40 mL/min OR serum creatinine ≤ 1.5 × ULN
   5. Total bilirubin ≤ 2.0 × ULN or ≤ 3.0 × ULN for subjects with Gilbert's syndrome
   6. AST, ALT, ALP ≤ 2.0 × ULN
6. Able and willing to comply with requested study visits and procedures.
7. Able and willing to provide written informed consent and HIPAA authorization

Exclusion Criteria:

1. Men and women (of reproductive potential) unwilling to use birth control and women who are pregnant or breastfeeding
2. Patient has primarily "diffuse" type AA (characterized by diffuse hair shedding)
3. Presence of another form of alopecia
4. Prior use of any of the following treatments: a. Aldesleukin b. Investigational IL-2 analog
5. Concurrent use of oral or topical treatments targeting hair growth or hair restoration (including but not limited to finasteride, dutasteride, topical minoxidil or oral minoxidil) if discontinuation or dosage change is planned during the study period.
6. Prior use of phototherapy and any systemic immunosuppressant (systemic steroids, cyclosporin, methotrexate or any other immunosuppressive therapy) or immunomodulating biologic therapy (including but not limited to dupilumab, tralokinumab, lebrikizumab, nemolizumab, rocatinlimab, or daxdilimab, whether marketed or investigational) within 3 months prior to Screening.
7. Prior use of any B-cell depleting agents, whether marketed or investigational, including but not limited to rituximab, ocrelizumab, ofatumumab, or belimumab, within 6 months prior to Screening.
8. Known hypersensitivity or history of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in the study.
9. History of diabetes mellitus, regardless of whether it is controlled or not.
10. History of myocardial infarction, congestive heart failure, uncontrolled arrhythmias, cardiac revascularization, stroke, uncontrolled hypertension, or uncontrolled diabetes within 6 months prior to Screening.
11. Significant organ dysfunction that is unstable or inadequately treated within 6 months prior to Screening.
12. History of cancer or lymphoproliferative disease, except for the following: adequately treated basal cell or squamous cell skin cancer without current evidence of disease.
13. Currently receiving any chronic systemic (oral or intravenous) anti-infective therapy for chronic infection (such as pneumocystis, cytomegalovirus, herpes zoster, or atypical mycobacteria).
14. Active tuberculosis (TB) (based on TB blood test or a TB skin test) or a history of inadequately treated TB.
15. Herpes zoster or cytomegalovirus (CMV) that resolved less than 2 months prior to Screening. Subjects with a history of frequent outbreaks of Herpes Simplex Virus (defined as 4 or more outbreaks a year).
16. Major surgery within 3 months prior to Screening visit or has a major surgery planned during the study.
17. Active systemic infection requiring parenteral antibiotic/antiviral therapy. All prior infections must have resolved following optimal therapy.
18. Prior organ allograft or allogeneic transplantation.
19. Positive based on serological screening for human immunodeficiency virus (HIV), hepatitis B or hepatitis C at screening.
20. Any ongoing toxicity from prior therapies that, in the judgment of the Investigator, may interfere with study treatment. All toxicities attributed to prior therapy must resolve to grade 1 or baseline before administration of the study treatment.
21. Psychiatric illness/social situations that would limit compliance with study requirements.
22. Other skin conditions that would interfere with study assessments of AA.
23. Other illness or a medical issue that in the opinion of the Investigator would exclude the subject from participating in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-16 (Actual); Primary Completion 2026-07-16 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) in Subjects Receiving HCW9302 Monotherapy | 9 Weeks
  Evaluate the safety profile of HCW9302 monotherapy in subjects with Alopecia Areata (AA), based on the incidence, type, and severity of adverse events (AEs) classified according to MedDRA.
Designate the recommended Phase 2 dose level (RP2D) for Phase 2 study of HCW9302 in subjects with AA | 9 Weeks

SECONDARY OUTCOMES:
Determine the percent change from baseline of Severity of Alopecia Tool (SALT) score (0-100) at Day 29 and Week 9 in AA subjects receiving HCW9302 | 9 Weeks
  A SALT score of 0 indicates no hair loss, while a score of 100 signifies complete hair loss.
Determine the change from baseline of Alopecia Areata-Investigator Global Assessment (AA-IGA) score at Day 29 and Week 9 in AA subjects receiving HCW9302 | 9 Weeks
  The AA-IGA contains 5 categories: 0 = None (SALT score of 0%); 1 = Limited (SALT score of 1% - 20%); 2 = Moderate (SALT score of 21% - 49%); 3 = Severe (SALT score of 50% - 94%); and 4 = Very Severe (SALT score of 95% - 100%).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - James A. Haley Veterans' Hospital, Tampa, Florida
  - The Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No